CLINICAL TRIAL: NCT05150002
Title: Cervical Spinal Cord Stimulation in Patients With Cerebral Vasospasm After Subarachnoid Haemorrhage: VasoStim Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor left
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VasoStim
Record Dates: First submitted 2021-11-15; First posted 2021-12-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Cerebral Vasospasm; Subarachnoid Hemorrhage
MeSH Terms: conditions — Vasospasm, Intracranial; Subarachnoid Hemorrhage | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cervical spinal cord stimulation on cerebral vasospasm after aneurysmal SAH (Experimental): Cervical spinal cord stimulation on cerebral vasospasm after aneurysmal SAH
  Interventions: Device: Spinal cord stimulation

INTERVENTIONS:
Device: Spinal cord stimulation — Cervical spinal cord stimulation on cerebral vasospasm after aneurysmal SAH

SUMMARY:
Cerebral vasospasm is characterized by a vasoconstriction of cerebral arteries causing a reduction of cerebral blood flow (CBF) and leading to ischemia and infarction of the brain parenchyma. Cerebral vasospasm is a serious complication of aneurysmal subarachnoid hemorrhage (SAH) with high morbidity and overall mortality of 40-50%.

Although the exact mechanisms of spinal cord stimulation (SCS) on the innervation of cerebral vessels are still unclear, several hypotheses have been formulated and studies in animals and human performed with very promising results.

This is a proof of concept study to better understand the effect and mechanisms of cervical spinal cord stimulation on cerebral vasospasm after aneurysmal SAH in human.

DETAILED DESCRIPTION:
Cerebral vasospasm is characterized by a vasoconstriction of cerebral arteries causing a reduction of cerebral blood flow (CBF) and leading to ischemia and infarction of the brain parenchyma. Cerebral vasospasm is a serious complication of aneurysmal subarachnoid hemorrhage (SAH) with high morbidity and overall mortality of 40-50%. The exact pathophysiological mechanisms underlying cerebral vasospasm are still not known in detail.

A wide range of different therapeutic options with various efficacies are available, triple-H therapy and endovascular treatment options like intra-arterial application of vasodilators e.g. Nimodipine or Papaverine or transluminal balloon angioplasty have been reported and are applied to prevent and treat cerebral vasospasm after SAH. Calcium channel blockers such as nimodipine or nicardipine improve outcome in patients after SAH and reduce the risk of secondary ischemia. The benefit of the different therapies is undoubted, but there is still potential for improvement concerning the rate of morbidity and mortality.

Although the exact mechanisms of spinal cord stimulation (SCS) on the innervation of cerebral vessels are still unclear, several hypotheses have been formulated and studies in animals and human performed with very promising results.

This is a proof of concept study to better understand the effect and mechanisms of cervical spinal cord stimulation on cerebral vasospasm after aneurysmal SAH in human.

Subjects are enrolled into the study, if radiographical vasospasms are detected in CTA, CTP, cerebral angiography or TCD.

SCS leads are implanted within 12h after study enrolment following the investigator's standard practice. SCS will be continuously delivered until day 14 after SAH. Doppler ultrasound is performed before SCS lead implantation and repeated after implantation on a daily basis and appearance of a new neurological deficit device until 24h after stopping the stimulation. Efficacy of cervical SCS is further evaluated by CTA or angiography and CTA/P performed 48h and 96h after lead implantation, as well as on day 14 after SAH before stopping the stimulation. The SCS electrode(s) are explanted on day 15. Intracerebral pressure is monitored from day 7-15. Headache, measured as NRS 0-10 and the consumption of analgesics are monitored from day 7-15, at discharge, at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Fisher 3 grade subarachnoid hemorrhage at presentation
* Secured aneurysm by clipping or coiling
* Is 18-75 years of age at the time of enrollment
* Cerebral vasospasm:

  * Cerebral angiography

    o Narrowing of vessel lumen > 66%
  * Transcranial Doppler ultrasound

    * Mean flow velocity > 150 cm/s or
    * Lindegaard Index > 3 or
    * increase > 50 cm/s within 24 hours
  * Intracranial CT angiography

    o Narrowing of vessel lumen > 66%
  * Intracranial CT perfusion o Time To Drain (TTD) > 4.7 seconds
* Is willing and capable of providing informed consent or existence of the presumed will of the patient by a relative or a legal representative
* Written confirmation by a study independent physician to guarantee patient interest
* Is willing and capable of complying with the study related requirements, procedures, and visits
* No findings on spinal imaging preventing SCS lead implantation
* Negative pregnancy test
* No breast feeding

Exclusion Criteria:

* Untreated ruptured aneurysm
* Cerebral infarction in the territory of the spastic arteries or massive disseminated infarction
* Signs of cerebral herniation
* Uncontrollable intracranial pressure
* Infection
* Coagulation disorder
* Is participating in another interventional trial
* Circulatory instability
* Severe congestive heart failure
* Patients with an elevated risk of bleeding
* Known allergy to implanted materials (Silicon, Titanium)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-06-30 (Actual); Primary Completion 2025-12-12 (Actual); Study Completion 2026-01-06 (Actual)

PRIMARY OUTCOMES:
Change of baseline flow velocity | 14 days after onset vasospasm
  The change of baseline flow velocity from the onset of vasospasm to day 14 assessed with Doppler ultrasound showing the effect of cervical SCS.

SECONDARY OUTCOMES:
Vasospasm changes in angiography and perfusion in CTP | 48 hours after stimulation
  Vasospasm changes in angiography and perfusion in CTP
Vasospasm changes in CTA and perfusion in CTP | 48 hours after stimulation
  Vasospasm changes in CTA and perfusion in CTP
Vasospasm changes in angiography and perfusion in CTP | 96 hours after stimulation
  Vasospasm changes in angiography and perfusion in CTP
Vasospasm changes in CTA and perfusion in CTP | 96 hours after stimulation
  Vasospasm changes in CTA and perfusion in CTP
Vasospasm changes in CTA and perfusion in CTP | 14 days after stimulation
  Vasospasm changes in CTA and perfusion in CTP
Vasospasm changes in angiography and perfusion in CTP | 14 days after stimulation
  Vasospasm changes in angiography and perfusion in CTP
Triple-H therapy | 14 days after stimulation
  Development of symptomatic vasospasm from onset to day 14 with need for Triple-H therapy
Angioplasty or intra-arterial application of vasodilators | 14 days after stimulation
  Development of symptomatic vasospasm from onset to day 14 with need for angioplasty or intra-arterial application of vasodilators
Intracerebral pressure (ICP) | Day 7- 14
  Intracerebral pressure (ICP)
Headache | Day 7- 14
  Headache measured by VAS Scale (Score 0-10 with 0 representing no pain, and 10 maximum pain intensity)
Consumption of analgesics | Day 7- 14
  Consumption of analgesics
Side effects of SCS | Day 7- 14
  Side effects of SCS

CONTACTS AND LOCATIONS:
Overall Officials: Janine Ai Schlaeppi, MD, Principal Investigator — Department of Neurosurgery, Inselspital
Locations (1):
- Dep. of Neurosurgery, Bern University Hospital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No